CLINICAL TRIAL: NCT00634335
Title: Echocardiographic Characteristics of High Endurance Israeli Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Dr. Sergio kobal, Soroka medical center
Other Study IDs: sor465808ctil
Record Dates: First submitted 2008-03-04; First posted 2008-03-13 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-02

CONDITIONS: Athlete's Heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- sk: professional Israeli bicyclists

SUMMARY:
The purpose of this study is to characterize the cardiac adaptive changes of professional Israeli bicyclists by using echocardiography.

DETAILED DESCRIPTION:
Adaptive cardiac changes, such as enlargement of left ventricle mass and enlargement of left ventricular wall was observed in athletes. The physiological limit of remodeling changes in accordance to sex, type of activity, intensity of activity, genetics and race.

Although many studies were conducted on this subject, it is still impossible to predict if an athlete from a certain sport will develop cardiac changes and their what will those changes characteristics will be.

Sudden cardiac death is the leading cause of death among young athletes, this is because of high physical activity in the presence of a hidden heart disease, therefore there is much debate about the needed screening tests for athletes.

In Israel, there is only one study in this subject that showed no significant cardiac changes in Olympic athletes of various types of sports. the study didn't focused on high endurance sport athletes such as professional bicyclists although cardiac endurance is a main factor in cardiac changes.

ELIGIBILITY:
Inclusion Criteria:

* Known athletes of the bicyclists organization of Israel or any other known organization for 2 year at least.
* Participated in at least one contest recognized by the bicyclists organization of Israel.
* Had been in training for the last 3 months at least, which included minimum of 8 hours a week in average

Exclusion Criteria:

* Do not suffer any known cardiac disease
* Had declared that they are not using drugs which are forbidden by the Olympic committee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: professional bicyclists in Israel
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Kobal, MD, Principal Investigator — Soroka medical center, Israel
Locations (1):
- Soroka University Medical Center, Beersheba, Israel